CLINICAL TRIAL: NCT07257068
Title: Checkpoint Inhibitor Associated Diabetes Mellitus: Early Recognition and Treatment (CERT) Project: A Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1541; NCI-2025-08623 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-11-18; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Checkpoint Inhibitor; Pilot Study; Diabetes Melletus
MeSH Terms: interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pilot Study Treatment wiith Infliximab (Experimental)
  Interventions: Other: Infliximab

INTERVENTIONS:
Other: Infliximab — Given by IV

SUMMARY:
To find out if taking a drug called infliximab (the "study drug") is safe and effective in reversing insulin dependence in CIADM.

DETAILED DESCRIPTION:
Primary Objective

1. To estimate the efficacy of infliximab in reversing insulin dependence in CIADM.

Secondary Objective

1. To evaluate the safety of infliximab when used for CIADM.
2. To estimate the duration of time off insulin for patients who are able to discontinue insulin.

ELIGIBILITY:
Eligibility Criteria

* Participants on ICI referred to endocrine for new diagnosis of CIADM, will be included provided they are within 12 months of last dose of ICI and if they have:

  * New onset diabetes≥ 200 mg/dl and/or A1c ≥6.5 OR
  * Worsening glycemic control: requiring insulin per clinician assessment (fasting glucose or average glucose on CGM>20% and /or A1c >0.5% from prior to ICI use ) AND /OR
  * If Presenting with DKA/HHS: include if within 6 weeks of presentation AND
  * Must have detectable random c-peptide level 0.2 - 1 ng/mL with blood glucose of 145 mg/dl
* Age ≥18 years. Because adverse event data are currently available on the use of infliximab in combination within participants <18 years of age, children are excluded from this study.
* ECOG performance status ≤2 (Karnofsky ≥60%,).
* Participants must have adequate organ and marrow function as defined below:

absolute neutrophil count ≥1,000/mcL platelets ≥100,000/mcL total bilirubin ≤ institutional upper limit of normal (ULN) AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN creatinine ≤ institutional ULN

Cardiac ejection fraction > 50%

* Participants with a prior or concurrent malignancy whose natural history or treatment does not interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of infliximab administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Participants already on insulin for pre-existing type 1 or type 2 diabetes.
* Participants with undetectable c-peptide levels i.e. <0.2 with blood glucose of 145 mg/dl or higher.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Participants with a h/o active TB or latent TB will be excluded.
* Participants with known history of any NYHA class heart failure or ejection fraction <50% will be excluded.
* Participants requiring supraphysiological doses of steroids i.e. prednisone >10mg of equivalent at the time of study entry, will be excluded
* Participants who have ICI hepatitis and myocarditis will be excluded
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities ≥ Grade 2) with the exception of alopecia.
* Participants who are receiving any other investigational agents for CIADM.
* History of allergic reactions or hypersensitivity attributed to compounds of similar chemical or biologic composition to Infliximab or other agents used in study.
* Required: any concomitant drugs used as defined in section 5.7 will be excluded.
* Participants with uncontrolled intercurrent illness: active infection/ sepsis
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and breastfeeding women are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with infliximab. Breastfeeding should be discontinued if the mother is treated with infliximab. These potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-04-14 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs). | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka C Iyer, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org